CLINICAL TRIAL: NCT06372652
Title: A Randomized, Double-blinded, Placebo-controlled Phase 1 Study of a Single Dose of a Subcutaneous Ultra-Long-Acting Somatostatin Analog (TE-8214 Solution) to Investigate the Safety, Tolerability, and Pharmacokinetics in Healthy Volunteers
Brief Title: A Phase 1 Study of TE-8214 Solution in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immunwork, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: TE-8214-001
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SAD Cohort (Experimental): Each participant will receive TE-8214 administered by subcutaneous injection across 5 Cohorts (Cohort 5 optional)
  Interventions: Drug: TE-8214 - SAD
- Placebo (Experimental): Each participant will receive matching volume doses of Placebo administered by subcutaneous injection
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TE-8214 - SAD — Cohort 1 - Single subcutaneous dose of 0.6 mg Cohort 2- Single subcutaneous dose of 1.2 mg Cohort 3 - Single subcutaneous dose of 2.0 mg Cohort 4 - Single subcutaneous dose of 3.0 mg or 4.0 mg Cohort 5 (Optional) - Single subcutaneous dose of 6.0 mg
  Arms: SAD Cohort
Drug: Placebo — Single subcutaneous dose of matching placebo across the cohorts
  Arms: Placebo

SUMMARY:
This is a Phase 1, first-in-human, randomized, double-blinded, placebo-controlled study to evaluate the safety, tolerability, and PK of TE-8214 in healthy volunteers. The study will assess single ascending doses (SAD) of TE-8214.

DETAILED DESCRIPTION:
This study will enroll approximately 32 eligible healthy volunteers.

The main purpose of this study is to evaluate the safety, tolerability, and PK of single ascending doses (SAD) of TE-8214. This study will involve 4 groups (called Cohorts) of 8 participants at a time, with each group receiving a higher dose than the group before. A further 8 participants may be randomized into an optional cohort.

Each participant will receive 1 dose of TE-8214 solution or placebo in a randomized, double-blinded manner and the IP will be administered by subcutaneous injection into the abdomen. For each cohort, there will be a sentinel group and a main group. In the sentinel group, 2 participants will be randomized to TE-8214 or placebo at a ratio of 1:1. if there are no safety concerns this will be followed by the main group dosing at the discretion of the investigator.

The total duration of the study for each participant is up to 16 weeks which consists of 28 days for Screening, confinement period of 3 days with dosing on Day 1 and a follow up period until Day 84.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, between 18 and 64 years old (inclusive, at the time of informed consent).
2. In good general health, as determined by past medical history, physical examination, vital signs, ECG, and laboratory tests at Screening and/or before the administration of IP at the discretion of the PI or designee.
3. Sign informed consent forms which include an explanation of the nature of the study, and the expected compliance with the requirements and restrictions of the study.

Exclusion Criteria:

1. Any abnormal laboratory values at Screening that are considered clinically significant by the PI or designee, or evidence of clinically significant abnormal findings at the physical examination at Screening, or significant illness within 2 weeks prior to dosing.
2. Have known allergies to octreotide, somatostatin analogs, or related compounds.
3. Have abnormal ECG findings at Screening that are considered by the PI or designee to be clinically significant, including, but not limited to: PR interval > 220 ms, QTcF > 450 ms (males) or > 470 ms (females), and/or arrythmias.
4. History of clinically significant allergy (including anaphylaxis), history or clinical evidence of pancreatic injury or pancreatitis.
5. History of gallstones, prior cholecystectomy is not exclusionary.
6. History of B12 deficiency.
7. History of hypothyroidism, or TSH > 4 mIU/L at Screening.
8. Any individual with a known history of diabetes mellitus, or HbA1c ≥ 6.5% at Screening. Individuals with previous gestational diabetes are eligible to participate, provided they do not currently have diabetes.
9. Women of childbearing potential (WOCBP) must be non-pregnant and must use an acceptable, highly effective double contraception from Screening until study completion.
10. Males must use an acceptable, highly effective double contraception from Screening until study completion and must not donate sperm until at least 90 days after the last dose of study drug.
11. Anything that the PI considers that would jeopardize the safety of the participant, prevent complete participation in the study, or compromise interpretation of study data.
12. Any skin condition and/or tattoo that may interfere with the evaluation of safety at the injection site.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-12-06 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of TE-8214 by the incidence of treatment-emergent adverse events (TEAEs) | From administration of IP on Day 1 until the EOS/ET visit (Day 84) post dose
Safety and tolerability of TE-8214 by the incidence of treatment-related adverse events | From screening until the EOS/ET visit (Day 84) post dose
Safety and tolerability of TE-8214 by the incidence of injection site reactions (ISRs) | On Day 1, 0 hour, 6 hours, 12 hours, 24 hours, 48 hours,72 hours, 96 hours, 168 hours post dose
Safety and tolerability of TE-8214 by the incidence of clinically significant laboratory findings | From Screening until EOS/ET (Day 84) post dose
Safety and tolerability of TE-8214 by the changes in physical examination findings | At Screening, Day -1, Day 2, Day 8, Day 28, Day 56, Day 84 post dose
Safety and tolerability of TE-8214 by the changes in ECG findings | At Screening, Day -1, Day 1, Day 2, Day 4, Day 8, Day 14, Day 28, Day 56, Day 84 post dose

SECONDARY OUTCOMES:
PK Parameters: Maximum observed concentration (Cmax) | On Day 1, Day 2, Day 3, Day 4, Day 5, Day 8, Day 10, Day 14, Day 21, Day 28, Day 56, Day 84 post dose
PK Parameters: Time to maximum observed concentration (Tmax) | On Day 1, Day 2, Day 3, Day 4, Day 5, Day 8, Day 10, Day 14, Day 21, Day 28, Day 56, Day 84 post dose
PK Parameters: Area under the concentration-time curve (AUC) from time zero to the last measurable concentration (AUC 0-last) | On Day 1, Day 2, Day 3, Day 4, Day 5, Day 8, Day 10, Day 14, Day 21, Day 28, Day 56, Day 84 post dose

CONTACTS AND LOCATIONS:
Locations (1):
- CMAX Clinical Research, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No